Official Title: Building mental health resilience in the COVID-19 pandemic.

**Brief Title:** Brief Video Interventions for Depression

NCT Number: NCT04643964

**Date of Document:** 8/30/2022

## Statistical Analysis Plan

Data were analyzed using SAS 9.4. Participants who failed one or more attention checks (e.g., "What is 124 + 1?") were excluded from analyses. We tested for possible condition differences between the entrée (i.e., an intervention focused on teaching participants one coping skill), sampler (i.e., an intervention providing an introduction to three coping skills), and no-intervention control conditions in depressive symptoms, coping skills, loneliness, age, and gender. We also evaluated whether there were condition differences in credibility or expectancy following the intervention.

To test the primary hypotheses, we evaluated potential condition differences in each outcome variable (viz., depressive symptoms, coping skills frequency, coping skill quality, and loneliness) at Time 2, controlling for the Time 1 level of that same variable. Baseline depressive symptoms were also included as a covariate in all models. Other covariates considered in these models were age, gender, and COVID interference. Covariates that were significant at p < .05were included in primary models. The only significant covariate identified was gender, which was limited to models examining coping skill frequency. The entrée condition's three separate interventions (cognitive skills, behavioral skills, or interpersonal skills) were combined for these analyses. In analyses of the coping skill frequency scale (the SERQ), repeated-measures regression with an unstructured covariance matrix was used to model the three subscales of interest (Cognitive, Behavioral, and Interpersonal) as repeated measures reflecting CBT skills. A variable indicating which skill was targeted in the assigned intervention was also included in the model. For instance, participants in the behavioral entrée had a score of '1' for the line reflecting the behavioral subscale and a '0' for the cognitive and interpersonal subscales. Participants in the sampler condition had scores of '1' for all three subscales.

In exploratory analyses, we conducted other specific comparisons of interest. These analyses included: comparing the entrée and sampler conditions without including the control condition and comparing each of the entrée variations with each other. We examined condition differences in risk of dropout using logistic regression. We also used logistic regression to examine condition differences in completing coping skill worksheets. Finally, we evaluated two potential moderators of any entrée versus sampler difference in outcomes: initial depression severity and preference for using one vs. multiple skills. We did not correct for multiple comparisons.